CLINICAL TRIAL: NCT01921153
Title: Encouraging Healthy Food Choices With an Environmental Intervention in Military Dining Facilities
Brief Title: An Environmental Intervention to Encourage Healthy Food Choices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United States Army Research Institute of Environmental Medicine (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 13-14H
Record Dates: First submitted 2013-07-31; First posted 2013-08-13 (Estimated); Last update posted 2016-05-04 (Estimated); Status verified 2016-05

CONDITIONS: Dietary Habits; Health Knowledge, Attitudes, Practice
MeSH Terms: conditions — Feeding Behavior; Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Short Intervention (Experimental): All participants will be measured for (1) baseline, (2) two-week environmental intervention: Healthy meal plates and trays, and (3) withdraw of intervention.
  Interventions: Other: Healthy meal plates and trays
- Long Intervention (Experimental): All participants will be measured for (1) baseline, (2) four-week environmental intervention: Healthy meal plates and trays, and (3) withdraw of intervention.
  Interventions: Other: Healthy meal plates and trays

INTERVENTIONS:
Other: Healthy meal plates and trays — The healthy meal plates and trays provide guidance for how to construct a meal in the military dining facility.

SUMMARY:
The primary objective of this study is to test effectiveness of an environmental intervention designed to encourage healthy food intake during meals. It is hypothesized that fruit, vegetable, whole grain, lean protein, and low-fat dairy consumption will increase during the intervention. It is also hypothesized that nutrition knowledge, attitudes, and behaviors will change as a result of the intervention. The findings from this study will provide insight into the applicability of this intervention in military dining facilities.

DETAILED DESCRIPTION:
Previous studies attempting to increase consumption of healthy foods in military dining facilities have had mixed results, and alternative approaches need to be considered. The present intervention was designed with the results of previous studies in mind, and as such, does not focus on labeling only healthy food choices. Instead, the present intervention aims to encourage consumption of nutritionally well-balanced meals using an environmental cue in military dining facilities.

ELIGIBILITY:
Inclusion Criteria:

* Military member or government civilian employee
* Normally eat in military dining facility at least 1 day per week.

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2013-08; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Change in dietary intake | Participants will be followed for 6-12 weeks
  Dietary intake will be assessed at lunches eaten in military dining facilities using the food photography method. The change in dietary intake from baseline to intervention will be assessed.

SECONDARY OUTCOMES:
Change in nutrition knowledge | Measured at beginning and end of the 6-12 week study.
  Nutrition knowledge specific to the intervention will be assessed with an experimenter-developed questionnaire.
Change in nutrition attitudes and behaviors (composite) | Measured at the beginning and end of the 6-12 week study.
  Nutrition attitudes and behaviors will be measured with a single composite experimenter-developed questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Tracey J Smith, PhD, Principal Investigator — United States Army Research Institute of Environmental Medicine
Locations (1):
- Natick Soldier Systems Center Dining Facility, Natick, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided